CLINICAL TRIAL: NCT06460506
Title: A Phase 3, Open-label Study Evaluating the Long-term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects 12 Months of Age and Older
Brief Title: Evaluation of Long-term Safety and Efficacy of ELX/TEZ/IVA in Cystic Fibrosis Participants 12 Months of Age and Older
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX22-445-123; 2023-509563-24-00 (Other: EU CT Number)
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Participants will receive ELX/TEZ/IVA in the morning and IVA in the evening.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination granules for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Granules for oral administration
  Other Names: VX-770; ivacaftor

SUMMARY:
The purpose of the study is to evaluate the long-term safety, tolerability, efficacy, and pharmacodynamics (PD) of elexacaftor (ELX)/tezacaftor (TEZ)/ivacaftor (IVA).

ELIGIBILITY:
Key Inclusion Criteria:

* Completed study drug treatment in the parent study VX22-445-122 Part B (NCT05882357) OR had study drug interruption(s) in the parent study but did not permanently discontinue study drug and completed study visits up to the last scheduled visit of the Treatment Period of the parent study

Key Exclusion Criteria:

* History of drug intolerance in the parent study that would pose an additional risk to the participant
* Current participation in an investigational drug trial other than the parent study

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Week 100

SECONDARY OUTCOMES:
Absolute Change in Sweat Chloride (SwCl) | From Baseline through Week 96

CONTACTS AND LOCATIONS:
Locations (18):
- Australia (3):
  - The Kids Research Institute Australia, Nedlands
  - The Royal Children's Hospital, Parkville
  - Queensland Children's Hospital, South Brisbane
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- Germany (3):
  - Charité Universitätsmedizin BerlinX, Berlin
  - Kinderklinik III, Abt. fur Pneumologie, Essen
  - Medizinische Hochschule Hannover, Hanover
- Erasmus Medical Center, Rotterdam, Netherlands
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Kinderspital Zurich, Zurich
- United Kingdom (6):
  - Children and Young Adults Research Unit, Cardiff
  - Leeds General Infirmary, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Children, London
  - Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing